CLINICAL TRIAL: NCT04984005
Title: The Interaction and Regulation Mechanism of Different Exercise Patterns With Metabolic Syndrome and Related Metabolic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M2021263
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: children and adolescents; Obesity; metabolic syndrome; overweight; exercise
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low intensity exercise training group (Experimental)
  Interventions: Behavioral: Low intensity exercise training
- Moderate intensity exercise training group (Experimental)
  Interventions: Behavioral: Moderate intensity exercise training
- Intermittent high intensity exercise training group (Experimental)
  Interventions: Behavioral: Intermittent high intensity exercise training

INTERVENTIONS:
Behavioral: Low intensity exercise training — The exercise method is broadcast gymnastics and sports dance. Through the design of different exercise intensities, This arm receives a low-intensity exercise training.
  Arms: Low intensity exercise training group
Behavioral: Moderate intensity exercise training — The exercise method is broadcast gymnastics and sports dance. Through the design of different exercise intensities, This arm receives a moderate-intensity exercise training.
  Arms: Moderate intensity exercise training group
Behavioral: Intermittent high intensity exercise training — The exercise method is broadcast gymnastics and sports dance. Through the design of different exercise intensities, This arm receives a high-intensity exercise training.
  Arms: Intermittent high intensity exercise training group

SUMMARY:
In order to obtain suitable exercise intervention model for children and adolescents with obese or metabolic syndrome in China, we conduct a RCT to examine the effects of different intensity exercise intervention on weight, and other cardiometabolic risk factors among children and adolescents, we also test the effects of exercise interventions on multi-omics such as metabolomics, gut microbiome, genetics, and explore the potential mechanisms by which exercise interventions modulate cardiometabolic risk. This is a randomized controlled study. Children and adolescents with obesity or metabolic syndrome were randomly divided into three groups, including low intensity exercise training group, moderate and intermittent high intensity exercise training group. The investigators will obtain organ hydrodynamics indexes by abdominal ultrasound and computational fluid dynamics technology, and obtain the metabolic regulation mechanism of the body in response to exercise through the detection of metabolism related small molecules in blood and urine and the analysis of intestinal flora, so as to explore the potential value and mechanism of different exercise modes in the treatment of obesity and metabolic syndrome. At the same time, the behavior and self-consciousness of children and adolescents will be investigated to obtain the suitable exercise intervention model for Chinese children and adolescents with obesity and metabolic syndrome. In conclusion, this study aims to demonstrate which exercise mode can alleviate obesity or reverse metabolic diseases, analyze which factors can sense exercise, and explore the potential mechanisms through mutil-omic approach, so as to improve metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of overweight or obesity or metabolic syndrome;
* Good academic performance in school;
* Willing to sign informed consent.

Exclusion Criteria:

* Clinical diagnosis of Cushing syndrome;
* Pathological obesity such as Prader-Willi syndrome and obesity caused by drug factors；
* Participated in other intervention studies within the previous three months;
* participant or their guardian has obvious intellectual or mental abnormalities.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 366 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline Obesity Indicators after 3 months of exercise | Before and after three months of exercise training
  BMI in kg/m^2
Changes from Baseline Body Fat Composition after 3 months of exercise | Before and after three months of exercise training
  Body fat composition (%)
Changes from Baseline Peak Metabolic Equivalent after 3 months of exercise | Before and after three months of exercise training
  Peak Metabolic Equivalent in MET
Changes from Baseline Blood Pressure after 3 months of exercise | Before and after three months of exercise training
  Blood pressure in mmHg
Changes from Baseline Fasting Blood Glucose after 3 months of exercise | Before and after three months of exercise training
  Fasting Blood Glucose in mmol/L
Changes from Baseline Total Serum Cholesterol after 3 months of exercise | Before and after three months of exercise training
  Total Serum Cholesterol in mmol/L
Changes from Baseline Triglyceride after 3 months of exercise | Before and after three months of exercise training
  Triglyceride in mmol/L
Changes from Baseline Serum High-density Lipoprotein Cholesterol after 3 months of exercise | Before and after three months of exercise training
  Serum High-density Lipoprotein Cholesterol in mmol/L
Changes from Baseline Serum Low-density Lipoprotein Cholesterol after 3 months of exercise | Before and after three months of exercise training
  Serum Low-density Lipoprotein Cholesterol in mmol/L
Changes from Baseline Sexual Hormones after 3 months of exercise | Before and after three months of exercise training
  Detection of hormone indicators related to growth and development

SECONDARY OUTCOMES:
Changes from Baseline Exercise Performance after 3 months of exercise | Before and after three months of exercise training
  VO2max/Kg in mL/min/Kg
Changes from Baseline Hepatic Hemodynamic Index after 3 months of exercise | Before and after three months of exercise training
  wall shear stress in proper hepatic artery，Pa
Changes from Baseline Bone Mineral Density after 3 months of exercise | Before and after three months of exercise training
  Using ultrasound bone density instruments for detection
Changes from Baseline C-reactive protein after 3 months of exercise | Before and after three months of exercise training
  Inflammatory Biomarker C-reactive protein in mg/L
Changes from Baseline Oxidative Stress Biomarkers after 3 months of exercise | Before and after three months of exercise training
  Oxidative Stress Biomarker MDA in nmol/mL
Changes from Baseline Serum Metabolomics after 3 months of exercise | Before and after three months of exercise training
  Metabolomics
Changes from Baseline Oral and Gut Microbiome after 3 months of exercise | Before and after three months of exercise training
  oral and gut microbiome
Changes from Baseline Viromics after 3 months of exercise | Before and after three months of exercise training
  viromics
Exome sequencing and genome sequencing | At baseline
  genetics
Changes from Baseline Proteomics after 3 months of exercise | Before and after three months of exercise training
  proteomics
Changes from Baseline Volatile Organic Compounds in Breath after 3 months of exercise | Before and after three months of exercise training
  Collect exhaled gas and use mass spectrometry for small molecule detection
Changes from Baseline Attention performance after 3 months of exercise | Before and after three months of exercise training
  Attention Survey Questionnaire
Changes from Baseline Sleep Quality after 3 months of exercise | Before and after three months of exercise training
  Wearing a heart rate monitoring watch to collect data
Changes from Baseline Total Thyroid Hormone after 3 months of exercise | Before and after three months of exercise training
  Total Thyroid Hormone in nmol/L
Changes from Baseline Liver steatosis after 3 months of exercise | Before and after three months of exercise training
  Abdominal ultrasound evaluation of the presence of hepatic steatosis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No